CLINICAL TRIAL: NCT03001505
Title: Registry to Evaluate Multi-modality Therapies for Pancreatic Cancer
Brief Title: Registry for Pancreatic Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Study design changed to clinical database only with no research question to be studied.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00075769
Record Dates: First submitted 2016-12-15; First posted 2016-12-23 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pancreatic cancer: Patients diagnosed with pancreatic cancer evaluated at this institution.

SUMMARY:
This is an observational, prospective and retrospective registry of patients with pancreatic cancer treated in Duke University Health System, which will examine patient and treatment effects on cancer outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer

Exclusion Criteria:

* Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pancreatic cancer who are treated at DUHS
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2037-04 (Estimated); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years
  Survival from Diagnosis to time of death

SECONDARY OUTCOMES:
Disease-free survival | 10 years
  length of time with no evidence of disease
Metastasis | 10 years
  Radiographic or surgical evidence of disease spread beyond the pancreas (or resection bed if post surgery).
Local recurrence | 10 years
  Radiographic evidence of disease recurrence in the resection bed, if post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sabino Zani, MD, Principal Investigator — DUHS
Locations (2):
- United States (2):
  - Duke University Health System, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No